CLINICAL TRIAL: NCT01370122
Title: The Prevalence and Predictive Factors of Pelvic Floor Disorders in Gynecologic Malignancy Survivors
Brief Title: Pelvic Floor Disorders in Survivors of Gynecologic Malignancies
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 35810
Record Dates: First submitted 2011-06-02; First posted 2011-06-09 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Uterine Cancer; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Cervical Cancer; Vulvar Cancer
Keywords: Women over the age of 20
MeSH Terms: conditions — Uterine Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects exposed to radiation
  Interventions: Other: Survey
- Subjects not exposed to radiation
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
Pelvic Floor dysfunction affects the quality of life of women. However, the prevalence and risk factors for pelvic floor disorders (PFD) in survivors of gynecologic malignancies are not known. The investigators plan to perform an observational study including survivors of gynecologic malignancies. Questionnaires for diagnosis of pelvic floor disorders will be mailed to survivors to generate prevalence rates and risk factors for PFD in women with a history of a gynecologic cancer diagnosis.

DETAILED DESCRIPTION:
Pelvic floor disorders negatively impact the quality of life of those afflicted by pelvic organ prolapse, lower urinary tract symptoms, defecatory or sexual dysfunction, or pain. Women who present for routine gynecologic care often have undiagnosed pelvic floor disorders, and physicians may not specifically question women to elicit pelvic floor symptoms. In the United States 24% of women report at least one pelvic floor disorder, which increases with age, parity , obesity. Gynecologic cancer survivors are a unique population who undergo a variety treatment regimens including surgery, chemotherapy, and radiation. Radical hysterectomy, a common surgical treatment for gynecologic cancers, is a well-established cause for lower urinary tract dysfunction. In contrast, data are lacking regarding risk factors for pelvic organ prolapse or fecal incontinence. Survivors of gynecologic malignancies may be at increased risk for symptomatic pelvic floor disorders, but may not be diagnosed due to lack of inquiry of these symptoms by practitioners. In addition, a recent qualitative study found that survivors of gynecologic malignancies believed that pelvic floor symptoms were an inevitable, untreatable corollary to treatment for their cancer and thus did not seek treatment. Furthermore, the study participants reported that they felt healthy despite these symptoms because of their oncologists assessment of their remission status. The lack of diagnosis and treatment of pelvic floor disorders has clinical and quality of life implications for the growing numbers of gynecologic malignancy survivors. The objective of this study is to identify the prevalence of an risk factors for pelvic floor disorders in women after treatment for gynecologic cancer. Our rationale for this project is that the investigators believe that pelvic floor disorders affect the quality of life of gynecologic cancer survivors and should be quantified. Successful completion of this study will provide evidence for practitioners to screen and treat pelvic floor disorders in gynecologic malignancy survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women with documented surgery for gynecologic malignancies at any of the three UPHS associated hospitals in center city Philadelphia (e.g., HUP, Pennsylvania hospital) and an accessible electronic medical record from the time of cancer diagnosis and beyond.
* Gynecologic cancer survivors at least 20 years of age diagnosed and treated for uterine, ovarian, peritoneal, fallopian tube, cervical, or vulvar tumors between 2008 to July 2010 will be included

Exclusion Criteria:

* Women who are pregnant, with benign tumors, those lost to follow-up, or deceased will be excluded from this study.
* Patients unable to complete a written survey due to physical or mental disabilities will also be excluded.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over the age of 20 with a history of uterine, ovarian, fallopian tube, peritoneal, cervical, or vulvar cancers.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence
  Urinary incontinence is the most common outcome of all symptomatic pelvic floor disorders in women

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States